CLINICAL TRIAL: NCT05744375
Title: Phase II Trial of TRAstuzumab deruxtecaN in firSt-line Treatment of HER2-positive Locally advanCEd or Metastatic Breast caNcer (MBC) Patients Considered Resistant to Trastuzumab + Pertuzumab + Taxane Due to Early Relapse."TRANSCENDER Study"
Brief Title: Trastuzumab Deruxtecan in First-line HER2-positive Locally Advanced/MBC Patients Resistant to Trastuzumab+Pertuzumab
Acronym: TRANSCENDER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped due to insufficient accrual (only two patients were included), and the sponsor has decided on its premature termination.
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2021-08; 2023-503627-26-00 (Other: EU CT Number)
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Trastuzumab deruxtecan; HER2-positive; Advanced Breast Cancer; Metastatic Breast Cancer; resistant to prior (neo) adjuvant anti-HER2 therapy.
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab deruxtecan (T-DXd) (Experimental): All patients enrolled will be treated with trastuzumab deruxtecan (T-DXd) 5.4 mg/kg IV every 3 weeks (± 3 days).
  The subject's weight at baseline will be used to calculate the initial dose. If during the course of treatment the subject's weight changes by ± 10% of the baseline weight, the subject's dose will be recalculated based on the subject's updated weight.
  Patients will receive T-DXd until unacceptable toxicity, progressive disease (PD), informed consent withdrawal, or other discontinuation criterion is met.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — All patients enrolled will be treated with trastuzumab deruxtecan (T-DXd) 5.4 mg/kg IV every 3 weeks (± 3 days).
  The subject's weight at baseline will be used to calculate the initial dose. If during the course of treatment the subject's weight changes by ± 10% of the baseline weight, the subject's dose will be recalculated based on the subject's updated weight.
  Patients will receive T-DXd until unacceptable toxicity, progressive disease (PD), informed consent withdrawal, or other discontinuation criterion is met.
  Other Names: Enhertu

SUMMARY:
The goal of this national, multicenter single arm phase II clinical trial is to study the efficacy, safety and tolerability of the administration of Trastuzumab Deruxtecan (T-DXd) in HER2-positive locally advanced or metastatic breast cancer (MBC) patients resistant to trastuzumab plus pertuzumab plus taxane due to early relapse.

The main questions it aims to answer are:

* To evaluate the antitumor activity of T-DXd in the first-line treatment of HER2-positive breast cancer patients resistant to trastuzumab-pertuzumab based therapy.
* To assess other efficacy measures.
* To evaluate safety and tolerability in all patients enrolled in the study.
* To evaluate health-related quality of life (HRQoL). Forty-one evaluable patients will be treated with trastuzumab deruxtecan (T-DXd) 5.4 mg/kg IV every 3 weeks (± 3 days). Patients will receive T-DXd until unacceptable toxicity, progressive disease, informed consent withdrawal, or other discontinuation criterion is met.

DETAILED DESCRIPTION:
This is a national, multicenter single arm phase II clinical trial to study the efficacy, safety and tolerability of the administration of Trastuzumab Deruxtecan (T-DXd) in HER2-positive locally advanced or MBC patients resistant to trastuzumab plus pertuzumab plus taxane due to early relapse.

Eligible patients will be enrolled and treated with T-DXd 5.4 mg/kg IV every 3 weeks.

The T-DXd dose will be recalculated in the event that patients experience body weight variations greater than 10% during the treatment period.

All patients enrolled will receive study therapy until radiographic or symptomatic progressive disease, unacceptable toxicity or withdraw of the informed consent, whatever occurs first.

Study population:

HER2-positive locally advanced or MBC patients who have not received prior chemotherapy or HER2 targeted therapy for advanced disease and with a Disease-Free Interval (DFI) of <12 months from the end of prior (neo)adjuvant anti-HER2 therapy.

Study Duration: The start date of the study is the date of the first site activation. Recruitment period will occur during approximately 24 months from the first patient in.

The end date of the study is the date of the last visit of the last patient (LPLV), including follow-up. The duration of the study will be approximately 68 months from the first patient in.

Performing exploratory objectives will be independent of the date of the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent obtained prior to any study-specific procedure.
2. Male or female patients of at least 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
4. Life expectancy ≥ 12 weeks.
5. Recurrent breast cancer that is unresectable locally advanced or metastatic.
6. Pathologically documented HER2-positive status by local laboratory determination, preferably on the most recent available Formalin-fixed paraffin-embedded (FFPE) tumor sample, according to the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) international guidelines valid at the time of the assay. In case of discordance in HER2 status in different biopsies, the result from the most recent biopsy will be used.
7. Pathologically documented Hormone Receptor (HR)-positive or -negative by local laboratory determination, preferably on the most recent available FFPE tumor sample, and according to ASCO/CAP international guidelines valid at the time of the assay. In case of discordance in HR status in different biopsies, the result from the most recent biopsy will be used.
8. Prior anti-HER2 based therapy (with trastuzumab plus pertuzumab plus taxane with or without trastuzumab-emtansine) in the (neo)adjuvant setting with a relapse while on therapy or within 12 months from the end of last anti-HER2 therapy.
9. Measurable disease assessed by the investigator based on RECIST version 1.1.
10. Left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
11. Adequate organ and marrow function defined as follows:

    1. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 (1.5x109/L).
    2. Platelet count ≥ 100,000/mm3 (100x109/L).
    3. Hemoglobin ≥ 9g/dL (90g/L).
    4. Creatinine clearance ≥ 30 mL/min as calculated using the standard method for the institution.
    5. Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN) if no liver metastases or < 3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
    6. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3.0 x ULN (< 5.0 × ULN in participants with liver metastases).
    7. Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5.0 x ULN if bone or liver metastases are present).
    8. Serum albumin ≥ 2.5 g/dL
12. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
14. Negative serum pregnancy test with a sensitivity of at least 25 milliInternational Units per milliliter of urine (mIU/mL) (unless permanent previous sterilization procedure such as bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) for premenopausal women, and for women who have experienced menopause onset < 12 months prior to first dose of therapy.

Exclusion Criteria:

1. Prior chemotherapy or HER2-targeted therapy for locally advanced or MBC (one prior endocrine therapy regimen for MBC without concurrent anti-HER2 therapy or radiotherapy is allowed).
2. Ineligible for treatment with T-DXd.
3. Any substance abuse or other medical conditions that, in the investigator's opinion, may interfere with patient's participation or study results.
4. Patients with spinal cord compression, leptomeningeal disease or clinically active central nervous system (CNS) metastases. Participants with clinically inactive brain metastases or treated brain metastases that are no longer symptomatic, and no needing corticosteroids or anticonvulsants may be enrolled in the study.
5. Active or prior documented interstitial lung disease (ILD)/pneumonitis or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
6. Lung criteria:

   1. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe Chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion etc.).
   2. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the electronic Case Report Form (eCRF) for patients who are enrolled in the study.
   3. Prior pneumonectomy.
7. Medical history of myocardial infarction within 6 months before registration, symptomatic congestive heart failure (CHF), troponin levels consistent with myocardial infarction as defined according to American College of Cardiologists (ACC) guidelines, unstable angina, or serious cardiac arrhythmia requiring treatment. QT interval corrected using Fridericia's formula (QTcF) > 470 msec (females) or > 450 msec (males) based on average of the screening triplicate 12-lead ECG.
8. History of active primary immunodeficiency, known Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).
9. Patients who received before treatment starts:

   1. Any investigational agent within 4 weeks.
   2. Chemotherapy within a period of time that is shorter than the cycle duration used for that treatment (e.g. < 3 weeks for fluorouracil, doxorubicine, epirubicin or < 1 week for weekly chemotherapy).
   3. Targeted therapy (e.g., antibodies): up to 4 weeks prior to starting study treatment.
   4. Endocrine therapy: tamoxifen or aromatase inhibitor within 2 weeks prior to starting study treatment.
   5. Radiotherapy within 2 weeks prior to starting study treatment. Patients who received prior radiotherapy to >25% of bone marrow are not eligible regardless of when it was administered.
   6. Major surgery or other anti-cancer therapy not previously specified within 4 weeks prior to starting study treatment.

   In any case, resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI-CTCAE version 5.0 grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion) is mandatory.Patients may be enrolled with chronic, stable grade 2 toxicities (defined as no worsening to > grade 2 for at least 3 months prior to enrollment and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as: chemotherapy-induced neuropathy or fatigue and immunotherapy-induced toxicities (e.g. endocrinopathies as hypothyroidism/hyperthyroidism, type 1 diabetes, hypoglycemia, adrenal insufficiency, adrenalitis and skin hypopigmentation [vitiligo]).
10. Have a diagnosis of any other malignancy within 3 years prior to inclusion, except for adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated and contralateral breast cancer.
11. Receipt of live, attenuated vaccine within 30 days prior to the first dose of T-DXd.
12. Prior treatment with T-DXd or allergic reaction to trastuzumab.
13. Patient is pregnant or breastfeeding or planning to become pregnant within the projected duration of the trial, starting at screening and through 7 months after the last dose of the study treatment. Male patients whose partners plan to become pregnant within the duration of the trial, starting at screening and through 4 months after the last dose of the study treatment.

    ✓ For premenopausal women it is necessary an agreement to remain complete abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study treatment.
    * Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include bilateral tubal litigation, male sterilization, and certain intrauterine devices (provided coils are copper banded).
    * Alternative, two methods (e.g. two barrier methods such as a condom and a cervical cap or combined with estrogen and progestogen) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.

    Female patients must not donate, or retrieve for their own use, ova from the time of enrollment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

    ✓ For men it is necessary an agreement to remain complete abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and to refrain from donating sperm during the same period, as defined below with female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of study treatment to avoid exposing the embryo.

    Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
14. Uncontrolled intercurrent illness including uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
15. Has substance abuse or any other medical/psychological conditions that may, in the opinion of the investigator, interfere with the patient's participation in the clinical study or evaluation of the clinical study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study treatment, and average of 18 months
  Objective Response Rate (ORR) is defined as the rate of complete response (CR) plus partial response (PR) based on the investigator's assessment using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1., out of the patients who received at least 1 dose of treatment (efficacy population).
  Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions.
  The ORR will be reported, including a 95% Confidence Interval (CI) using the Clopper-Pearson method.
  A sensitivity analysis will be performed using the Intent to treat population (ITT) population.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Through study treatment, and average of 18 months
  Progression-Free Survival (PFS) is defined as the time from the date of enrollment to the date of disease progression, based on the investigator's assessment using RECIST version 1.1., or death from any cause, whichever occurs first.
  PFS data will be censored on the date of the last tumor assessment on study for patients who do not have objective tumor progression and who have not died due to any cause while on study. Additionally, patients who start a new anti-cancer therapy prior to documented progression disease (PD) will be censored at the date of the last tumor assessment prior to the start of the new therapy. PD is defined using RECIST, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  PFS analysis will be performed in the safety population. PFS will be assessed using the Kaplan-Meier method. The median event time and 95% CI will be estimated if reached.
Overall Survival (OS) | Through study, and average of 36 months
  Overall Survival (OS) is defined as the time from the date of enrollment to the date of death from any cause.
  OS data will be censored on the last date the patient is known to be alive. OS analysis will be performed in the safety population. OS will be assessed using the Kaplan-Meier method. The median event time and 95% CI will be estimated if reached.
Time to treatment response (TTR) | Through study treatment, and average of 18 months
  Time to treatment response (TTR) is defined as the time from the date of enrollment to the date of first documentation of objective tumor response (CR or PR).
  TTR analysis will be performed in the efficacy population in patients with an Objective Response (OR).
  TTR will be assessed using the Kaplan-Meier method. The median event time and 95% CI will be estimated.
Duration of response (DoR) | Through study treatment, and average of 18 months
  Duration of response (DoR) is defined as the time from the date of first documentation of objective tumor response (CR or PR) to the date of first documented progressive disease based on the investigator's assessment using RECIST version 1.1., or death from any cause, whichever occurs first.
  DoR will be censored on the date of the last tumor assessment on study for patients who do not have objective tumor progression and who have not died due to any cause while on study. Additionally, patients who start a new anti-cancer therapy prior to documented PD will be censored at the date of the last tumor assessment prior to the start of the new therapy.
  DoR analysis will be performed in the efficacy population in patients with an OR.
  DoR will be estimated using Kaplan-Meier methods. The median event time and 95% CI will be estimated if reached.
The Number of Participants Who Experienced Adverse Events (AE) Related to Study Treatment | Through study treatment, and average of 18 months
  Safety assessments will be performed at baseline and during the study: Vital signs assessments (blood pressure, pulse and body temperature), measurement of left ventricular ejection fraction, triplicate 12-lead electrocardiogram, laboratory assessments (hemoglobin, White Blood Cell, Absolute Neutrophil Count, Lymphocytes, platelet count, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, total bilirubin, serum creatinine, creatinine clearance, sodium, potassium, total calcium, blood urea nitrogen (or urea), albumin, Troponin Test, Coagulation testing (International Normalized Ratio, activated partial thromboplastin time), pregnancy test , ophthalmologic assessments (visual acuity testing, slit lamp examination, fundoscopy), Viral serology.
  AEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
  The toxicity of study treatments will be evaluated in the safety population.
Changes from baseline in the global health status score (GHS) | Through study treatment, and average of 18 months
  Change from baseline in the GHS and each scale of the EORTC Quality of Life Questionnaire-Core 30 (QLQ-C30) will be presented at each scheduled time point for the GHS score and each of the functionals and symptoms scales from the QLQ-C30 questionnaires. Longitudinal analysis of scores will be performed using linear mixed models.
  QLQ-C30 is composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status/QoL scale, and 6 single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time to deterioration (TTD) in quality of life (QoL) | Through study treatment, and average of 18 months
  Time to deterioration (TTD) in QoL is defined as the time from the date of enrollment to the date of first detection of a deterioration event. A deterioration event is defined as an increase of ≥ minimally important difference (MID) from baseline for the EORTC QLQ-C30 symptom scales and a decrease of ≥ MID from baseline for the EORTC QLQ-C30 functional scales and GHS scale. It will be assessed using the Kaplan-Meier. Method. The median event time and 95% CI for the median will be estimated if reached. TTD will be censored at the date of the last QoL assessment prior to the start of a new therapy.

OTHER OUTCOMES:
Progression-Free Survival 2 (PFS2) | Through study, and average of 36 months
  PFS2 is defined as the time from the date of enrollment to the date of disease progression to the second line of therapy. PFS2 data will be censored on the last date in which the patient was known not to have tumor progression or death due to any cause within the second line of therapy. Additionally, patients who start a third line therapy prior to progression to the second line will be censored at the date of the start of the third line therapy.
  PFS2 will be performed in the safety population. PFS2 will be assessed using the Kaplan-Meier method. The median event time and 95% CI will be estimated if reached.
Progression-Free Survival 3 (PFS3) | Through study, and average of 36 months
  PFS3 is defined as the time from the date of enrollment to the date of disease progression to the third line of therapy. PFS2 data will be censored on the last date in which the patient was known not to have tumor progression or death due to any cause within the second line of therapy. Additionally, patients who start a third line therapy prior to progression to the second line will be censored at the date of the start of the third line therapy.
  PFS3 will be performed in the safety population. PFS3 will be assessed using the Kaplan-Meier method. The median event time and 95% CI will be estimated if reached.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — Hospital General Universitario Gregorio Marañón. Madrid, Spain.; Study Director Study Director, Study Director — Hospital del Mar. Barcelona, Spain.
Locations (19):
- Spain (19):
  - Hospital Universitario de Jeréz De La Frontera, Cadiz, Andalusia
  - Hospital Universitario de Jaén, Jaén, Andalusia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital San Juan de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org